CLINICAL TRIAL: NCT03586817
Title: COMPARATIVE STUDY BETWEEN PALONOSETRON AND FOSAPREPITANT IN THE PROFILAXIA OF POSTOPERATIVE NAUSEA AND VOMITING IN WOMEN SUBMITTED TO VIDEOLAPAROSCOPIC COLECISTECTOMIES
Brief Title: PALONOSETRON X FOSAPREPITANT IN PONV
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Federal de Bonsucesso (Other)
Responsible Party: Principal Investigator, Estevão Braga, Clinical Professor, Hospital Federal de Bonsucesso
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 89510518.6.0000.5253
Record Dates: First submitted 2018-06-29; First posted 2018-07-16 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Nausea and Vomiting, Postoperative
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Palonosetron; fosaprepitant

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Palonosetrona (Active Comparator): Palonosetron 75 mcg during the anesthesia
  Interventions: Drug: Palonosetron
- Fosaprepitant (Active Comparator): Fosaprepitant 150 mg during the anesthesia
  Interventions: Drug: Fosaprepitant

INTERVENTIONS:
Drug: Palonosetron — 75 mcg during the anesthesia
  Arms: Palonosetrona
Drug: Fosaprepitant — 150 mg during the anesthesia
  Arms: Fosaprepitant

SUMMARY:
Cholelithiasis (presence of gallbladder stones) is prevalent in 10 to 15% of the world population. This disease can lead to serious complications such as cholecystitis, cholangitis and pancreatitis. Video-laparoscopic cholecystectomy (CVL) is considered the gold standard treatment of this condition.

Despite ongoing research and development of new drugs and techniques, postoperative nausea and vomiting (PONV) are frequent, lead to unexpected hospitalizations, delay hospital discharge, increase hospital costs, and cause patient dissatisfaction. Video-laparoscopic surgeries are cited in the literature as a risk factor for PONV, with an incidence of up to 75% in cases where prophylactic drugs are not used.Through the simplified Apfel score, it is possible to determine the risk for PONV. This risk classification is based on four risk factors: female gender, non-smoking, postoperative use of opioids and previous history of PONV. The incidence of PONV would be 10%, 20%, 40%, 60% and 80%, respectively, if none, one, two, three or four risk factors are present.

Antiemetics recommended for prophylaxis of PONV in adults include 5-hydroxytryptamine (5-HT3) receptor antagonists (ondansetron, dolasetron, granisetron, tropisetron, ramosetron and palonosetron), neurokinin-1 (NK-1) receptor antagonists (aprepitant), (dendrohydrin and haloperidol), antihistamines (dimenhydrin and meclizine), and anticholinergics (scopolamine).

DETAILED DESCRIPTION:
The prospective, randomized and double-blind clinical trial will be performed at the Federal Hospital of Bonsucesso (HFB), Rio de Janeiro, RJ.

The Informed Consent Form (TCLE) will be presented and signed, on an outpatient basis, by each of the volunteer participants, who will be guided about the risks and benefits of the research, according to resolution CNS 466/12. A total of 100 female patients, aged between 18 and 60 years, ASA I and II, submitted to elective laparoscopic cholecystectomies, were randomly assigned to two groups: Group P (GP) will receive palonosetron 75 mcg and the other Group F GF), you will receive fosaprepitanto 150 mg. Palonosetron and fosaprepitanto are not standard medications in HFB. Both will be purchased and will be in the possession of the principal investigator, who undertakes to obey the current norms of the hospital institution and ensure the quality, storage and adequate stability of medications.

Patients will not receive preanesthetic medication. They will be monitored in the operating room with noninvasive blood pressure, electrocardioscopy, pulse oximetry, capnography, capnometry and bispectral index (BIS).

Patients will have a cannulated peripheral vein, be pre-oxygenated with oxygen at 100% for 5 minutes and anesthetic induction will be performed with intravenous administration (e.v.) of fentanyl 3 mcg / kg; lidocaine 1.5 mg / kg and propofol 2 mg / kg. Tracheal intubation will be facilitated after 3 minutes of administration of rocuronium 0.6 mg / kg e.v. After induction of anesthesia, the antiemetics, depending on the group studied, will be administered e.v. in solution containing 100 ml of 0.9% strength.

Maintenance of anesthesia will be with sevoflurane 2 L / min in 50% oxygen / air, with its concentration adjusted to maintain BIS between 40-60. Remifentanil 0.05 mcg / kg / min at 0.2 mcg / kg / min via e.v. may be given intraoperatively if the heart rate or blood pressure rises by more than 20% of the baseline values. Additional doses of rocuronium may also be given as needed. Patients will receive paracoxib 40 mg, dipyrone 50 mg / kg and ranitidine 50 mg e.v. after tracheal intubation. The surgical wound will be infiltrated with 20 ml of 0.5% ropivacaine before the sutures. The neuromuscular blockade will be reversed with neostigmine 0.04 mg / kg and atropine 0.02 mg / kg per e.v. Morphine 0.03 mg / kg e.v. will be given at the end of the surgery. The inflation of the pneumoperitoneum with CO2 (carbon dioxide), will have as limit abdominal pressure of 15 mmHg.

A physician not participating in the research will be aware of which antiemetic has been administered and will be responsible for the postoperative prescription of the patients. Both groups will have metoclopramide 10 mg e.v. as rescue medication for PONV.

For the purpose of the study, nausea will be defined as an unpleasant and involuntary sensation of vomiting, without the expulsion of stomach contents, and vomiting as expulsion of the stomach contents.

The patients will be visited by the research team 2, 6, 24 and 48 h after the end of the surgery, being questioned about the frequency and intensity of PONV, as well as other adverse effects. Researchers will not have access to prescription and medical records within the first 48 hours postoperatively.

After the last clinical evaluation, the researchers will analyze the prescription and note the use of morphine and rescue metoclopramide. They will also answer a question about the degree of satisfaction with the anti-emetic therapy used and will have 3 "Unsatisfied, satisfied or very satisfied" response options. Regarding the total cost of antiemetic therapy, it will be based on the ANVISA (National Health Surveillance Agency) table.

ELIGIBILITY:
Inclusion Criteria:

* women
* Non fumant
* cholelitiasis

Exclusion Criteria:

* severe heart, pulmonay, renal or liver diseases
* Tabagism

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Fenale
Enrollment: 100 (Estimated)
Dates: Start 2019-03-02 (Estimated); Primary Completion 2019-03-02 (Actual); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of complete responder | 48 hours
  individuals without nausea or vomiting

SECONDARY OUTCOMES:
Nausea | the first postoperative 48 hours
  questionnaire on the number of individual episodes of nausea
vomiting | the first postoperative 48 hours
  questionnaire on the number of individual episodes of vomiting

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Federal de Bonsucesso, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stinton LM, Shaffer EA. Epidemiology of gallbladder disease: cholelithiasis and cancer. Gut Liver. 2012 Apr;6(2):172-87. doi: 10.5009/gnl.2012.6.2.172. Epub 2012 Apr 17. PMID 22570746
- [Background] Chandrakantan A, Glass PS. Multimodal therapies for postoperative nausea and vomiting, and pain. Br J Anaesth. 2011 Dec;107 Suppl 1:i27-40. doi: 10.1093/bja/aer358. PMID 22156268
- [Background] Apfel CC, Roewer N. Risk assessment of postoperative nausea and vomiting. Int Anesthesiol Clin. 2003 Fall;41(4):13-32. doi: 10.1097/00004311-200341040-00004. No abstract available. PMID 14574212
- [Background] Muchatuta NA, Paech MJ. Management of postoperative nausea and vomiting: focus on palonosetron. Ther Clin Risk Manag. 2009 Feb;5(1):21-34. Epub 2009 Mar 26. PMID 19436621
- [Background] Singh PM, Borle A, Rewari V, Makkar JK, Trikha A, Sinha AC, Goudra B. Aprepitant for postoperative nausea and vomiting: a systematic review and meta-analysis. Postgrad Med J. 2016 Feb;92(1084):87-98. doi: 10.1136/postgradmedj-2015-133515. Epub 2015 Dec 1. PMID 26627976